CLINICAL TRIAL: NCT06549634
Title: Biomarkers of AKI in Patients With Multiple Myeloma Receiving Daratumumab: A Pilot Study
Brief Title: Biomarkers of AKI in Patients Receiving Daratumumab
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Shruti Gupta, Associate Physician, Director of Onconephrology, Brigham and Women's Hospital
Other Study IDs: 23-270
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Acute Kidney Injury; Multiple Myeloma; Light Chain Nephropathy
MeSH Terms: conditions — Acute Kidney Injury; Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10mL urine 5mL EDTA-plasma 5 mL serum Collections on day 0 and day 30
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with multiple myeloma: Patients with multiple myeloma being newly initiated on daratumumab
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab is not being administered as part of the study. Patients will receive daratumumab as part of their clinical care, and blood and urine will be collected in order to measure biomarkers pre- and post-daratumumab administration

SUMMARY:
The goal of this prospective observational study is to understand changes in urinary and blood biomarkers associated with acute kidney injury (AKI) in patients newly diagnosed with multiple myeloma and being treated with Daratumumab SC. The aims of the study are:

To measure changes in plasma and urinary biomarkers of AKI before initiation of Daratumumab therapy and 30 days after initiation of therapy.

To establish whether these biomarkers serve to aid in early detection and prevention of AKI

Participants will give urine and blood samples at their normally scheduled lab appointments.

DETAILED DESCRIPTION:
Serum creatinine is an insensitive marker of AKI, often rising late and after significant injury has already occurred. A number of novel markers have recently been shown to have utility in the early detection of AKI. These markers have shown promise in preclinical and human studies in multiple other clinical settings (e.g., cardiac surgery, coronary angiography, critical illness), but have not been studied in the context of multiple myeloma. Specifically, elevated pre-procedural plasma levels of soluble urokinase-type plasminogen activator receptor (suPAR), the circulating form of a membrane-bound protein expressed by immunologically active cells, have been demonstrated to be predictive of AKI patients undergoing coronary angiography, cardiac surgery, and in critically ill patients (Hayek et al., NEJM, 2020), and levels rise early after injury. Similarly, urinary levels of Dickkoph-3 (DKK3), a stress-induced tubular epithelia-derived glycoprotein, have been demonstrated to predict AKI after cardiac surgery and following administration of iodinated contrast (Schunk et al., Lancet, 2019).

The aim of this study is to conduct a pilot, prospective, non-interventional study testing changes in novel plasma and urinary biomarkers of kidney injury in patients with newly-diagnosed multiple myeloma treated with daratumumab who are at risk for AKI.

The hypothesis is that patients with multiple myeloma and at risk for developing AKI, but without AKI at baseline, will have at least a 10% decline in plasma soluble urokinase-type plasminogen activator receptor and urinary levels of Dickkoph-3 following treatment with daratumumab.

The primary outcome(s) will be changes in plasma suPAR and urinary levels of DKK3 between treatment initiation of daratumumab (day 0, or up to 7 days prior) and day +30 (+/-7 days) from the time of treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age
* Patients can be on a clinical trial
* Patients must have had a confirmed new diagnosis of MM following revised IMWG criteria

  1. New diagnosis of systemic multiple myeloma defined as no documented history of prior multiple myeloma.
  2. Further, no prior systemic treatment with anti-myeloma agent is permitted with the exception of corticosteroids for no more than 4 weeks.
  3. Prior history of receiving radiation therapy for the treatment of plasmacytoma or lytic lesions, is permitted on the study.
* Patients receiving SC daratumumab
* Patients must be able to sign the informed consent
* Patients must be at risk for AKI and meet at least two of the three following criteria: age ≥65; baseline eGFR <60; or use of NSAIDs (not including aspirin), bisphosphonates, intravenous contrast, diuretics, or RAS inhibitors in the 14 days preceding treatment initiation

Exclusion Criteria:

* End stage renal disease (e.g, on long-term dialysis or with a kidney transplant and on long-term dialysis) at the time of starting daratumumab
* Acute kidney injury defined as a ≥1.5-fold rise in baseline SCr, where baseline SCr is the lowest SCr in the 365 days preceding receipt of daratumumab, or with AKI on RRT
* Previous exposure to daratumumab or other anti-CD38 therapy
* Patients receiving intravenous daratumumab
* Exposure to concomitant chemotherapy which could be perceived as nephrotoxic within 30 days of receipt of daratumumab (e.g., cisplatin, mTOR inhibitors)
* Moribund patients (e.g., those expected to die in the next 30 days from the time of screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Plasma and Urine Biomarkers | 30 days
  The primary outcome(s) will be changes in plasma suPAR and urinary levels of DKK3 between treatment initiation of daratumumab (day 0, or up to 7 days prior) and day +30 (+/-7 days) from the time of treatment initiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States